CLINICAL TRIAL: NCT01482026
Title: Sensitivity of ADHD-IV Rating Scale in the Evaluation of the Evolution of Attention Disorders Associated With Childhood Epilepsy : a Validation Study
Brief Title: Attention-Deficit Hyperactivity Disorder (ADHD) Rating Scale and Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011.682/25
Record Dates: First submitted 2011-11-24; First posted 2011-11-30 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2016-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; Attention deficit; ADHD rating scale IV
MeSH Terms: conditions — Epilepsy; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treated patients (Experimental): Patients for whom ADHD treatment is introduced at enrolment. Evolution of the ADHD Rating Scale-IV inattention subscore
  Interventions: Other: ADHD Rating Scale-IV
- Non treated patients (Experimental): Patients for whom no ADHD treatment is required at enrolment. Evolution of the ADHD Rating Scale-IV inattention subscore
  Interventions: Other: ADHD Rating Scale-IV

INTERVENTIONS:
Other: ADHD Rating Scale-IV — ADHD Rating Scale-IV test
  Arms: Treated patients
Other: ADHD Rating Scale-IV — ADHD Rating Scale-IV test
  Arms: Non treated patients

SUMMARY:
The cognitive and psychiatric comorbidities are crucial endpoints in epileptic patients. Among these comorbidities, the Attention-Deficit Hyperactivity Disorder (ADHD) accounts for one of the most important in terms of frequency and psychosocial and educational consequences.

In these conditions, our study was designed to estimate the sensitivity to changes of the different sub-scores of the ADHD rating Scale IV (ADHD RS IV) in epileptic patient. This will then optimize our methodological approach for a therapeutic trial.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6 to 15 years and 11 months;
* male or female;
* with a diagnosis of ADHD : predominantly inattentive or combined hyperactive-impulsive and inattentive according to the DSM IV criteria;
* children who agreed to participate to the protocol and whose legal representatives have clearly expressed their non-opposition to participate.

Exclusion Criteria:

* Patients below 6 years old or patients older than 16 years;
* with a diagnosis of ADHD predominantly hyperactive-impulsive subtype ADHD according to the DSM IV criteria;
* mental retardation defined by a score < 70 at the verbal comprehension index and the perceptual reasoning score of the Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV)
* established diagnosis of any psychiatric co-morbidity other than ADHD according to the DSM IV criteria (pervasive developmental disorders including autism, bipolar disorder, psychotic disorder).

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evolution of the ADHD rating scale IV inattention subscore | Change from baseline in ADHD rating scale IV inattention subscore at 12 to16 weeks
  Evolution of the ADHD rating scale IV inattention subscore in treated versus non treated patients, after 12 to 16 weeks.

SECONDARY OUTCOMES:
Evolution of the ADHD rating scale IV global score | Change from baseline in ADHD rating scale IV global score at 12 to16 weeks
  Evolution of the ADHD rating scale IV global score in treated versus non treated patients, after 12 to 16 weeks.
Evolution of the ADHD rating scale IV hyperactivity subscore | Change from baseline in ADHD rating scale IV hyperactivity subscore at 12 to16 weeks
  Evolution of the ADHD rating scale IV hyperactivity subscore in treated versus non treated patients, after 12 to 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain RHEIMS, MD, Principal Investigator — Service de Neurologie Fonctionnelle et Epileptologie, Hôpital Neurologique Pierre Wertheimer, Hospices Civils de Lyon
Locations (15):
- France (15):
  - Service de Neurologie pédiatrique, CHU d'Amiens, Amiens
  - Service de Neurologie Pédiatrique, CHU d'Angers, Angers
  - Service de Neurologie pédiatrique, CHU de Besançon, Besançon
  - Unité de Neurologie de l'Enfant et de l'Adolescent, Hôpital Pellegrin, Bordeaux
  - Institut des Epilepsies de l'Enfant et de l'Adolescent, Hôpital Femme Mère Enfant, Bron
  - Service de Neurologie Fonctionnelle et Epileptologie, Hôpital Neurologique Pierre Wertheimer, Bron
  - Service d'épileptologie pédiatrique, CHR de Chambéry, Chambéry
  - Cabinet Médical du Dr ISNARD, Lyon
  - Service de Neurologie pédiatrique, Hôpital de la Timone, Marseille
  - Service de Neurologie Pédiatrique, Hôpital Robert-Debré, Paris
  - Service de Neurologie pédiatrique, Hôpital Neckert-Enfants malades, Paris
  - Service de Pédiatrie, Hôpital Sud, Rennes
  - Centre Référent des Epilepsies Rares, Hôpital de Hautepierre, Strasbourg
  - Service de Neurologie Pédiatrique, Hôpital des Enfants, Toulouse
  - Service de Neurologie Pédiatrique, CHU de Tours, Tours

REFERENCES:
- [Result] Mercier C, Roche S, Gaillard S, Kassai B, Arzimanoglou A, Herbillon V, Roy P, Rheims S. Partial validation of a French version of the ADHD-rating scale IV on a French population of children with ADHD and epilepsy. Factorial structure, reliability, and responsiveness. Epilepsy Behav. 2016 May;58:1-6. doi: 10.1016/j.yebeh.2016.02.016. Epub 2016 Mar 15. PMID 26991745